CLINICAL TRIAL: NCT07253389
Title: A Multicenter Randomized Controlled Trial: Comparison of Underdilated Versus Standard Transjugular Intrahepatic Portosystemic Shunt in Preventing Rebleeding From Esophagogastric Varices in Patients With Cirrhosis
Brief Title: Comparison of Underdilated Versus Standard TIPS in Preventing Variceal Rebleeding in Patients With Cirrhosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Tie Jun, Director of clinical research, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20252233-F-2
Record Dates: First submitted 2025-09-30; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Liver Cirrhosis; Gastroesophageal Varices Bleeding
Keywords: Liver Cirrhosis; Esophageal and gastric variceal bleeding; Transjugular intrahepatic portosystemic shunt; Hepatic encephalopathy
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy

STUDY DESIGN:
Intervention Model Description: This multicenter, single-blind randomized controlled trial (1:1 allocation) evaluates whether underdilated TIPS effectively controls variceal bleeding and reduces overt hepatic encephalopathy in cirrhotic patients. Conducted across 5 Chinese tertiary Grade A hospitals (Xijing Hospital as coordinating center), participants undergo pre-TIPS screening. Stratified block randomization ensures balance: stratified by center, then by sex, age (<60 vs. ≥60), Child-Pugh class (<9 vs. ≥9), bleeding indication (acute vs. secondary prophylaxis), variceal type (esophageal/GOV1 vs. GOV2/IGV1), and cirrhosis etiology (hepatitis B vs. non-hepatitis B). 85 patients per group are randomized to underdilated (experimental) or standard-diameter (control) TIPS.
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the nature of the interventions, investigators and procedural nursing staff were aware of group assignments. However, patients, follow-up researchers (responsible for data collection and endpoint assessment), and statisticians were blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard TIPS (Active Comparator): Standard TIPS Group: In the standard group, the TIPS stent will be progressively dilated (starting at 8 mm of diameter) to the minimum diameter needed to achieve a portosystemic pressure gradient (PSPG) below 12 mm Hg.
  Interventions: Procedure: Standard TIPS
- Underdilated TIPS (Experimental): Underdilated TIPS Group:In this group, the TIPS stent was underdilated using a 6-mm balloon, and the immediate post-procedure portal pressure gradient (PPG) was measured.
  Interventions: Procedure: Underdilated TIPS

INTERVENTIONS:
Procedure: Underdilated TIPS — The procedure will be performed via a transjugular approach, involving puncture from the hepatic vein or inferior vena cava into the portal venous system. Upon successful cannulation, direct portography will be performed to visualize varices and determine the optimal shunt tract, followed by targeted variceal embolization. A Novel VIATORR® Controlled Expansion (VCX) stent graft (W. L. Gore & Associates, Arizona, USA) will then be deployed intrahepatically to establish the shunt. Subsequently, a 6-mm balloon will be used for suboptimal expansion of the TIPS stent, and the immediate portosystemic pressure gradient (PPG) will be measured.
  Arms: Underdilated TIPS
Procedure: Standard TIPS — The procedure will be performed via a transjugular approach, with puncture conducted from the hepatic vein or inferior vena cava into the portal venous system. After successful cannulation, direct portography will be performed to visualize gastroesophageal varices and identify the optimal shunt tract, followed by targeted variceal embolization. A novel VIATORR® Controlled Expansion (VCX) stent graft (W. L. Gore & Associates, Arizona, USA) will then be deployed intrahepatically to establish the transjugular intrahepatic portosystemic shunt (TIPS). Subsequently, the TIPS stent will be progressively dilated (starting at 8 mm of diameter) to the minimum diameter needed to achieve a portosystemic pressure gradient (PSPG) below 12 mm Hg.
  Arms: Standard TIPS

SUMMARY:
Transjugular intrahepatic portosystemic shunt (TIPS) is a key therapeutic intervention for complications of portal hypertension. However, the risk of post-procedural hepatic encephalopathy (HE) limits its broader clinical application. In the management of gastroesophageal variceal bleeding, the primary goal of TIPS is to reduce the portosystemic pressure gradient (PPG) to less than 12 mmHg (16 cmH₂O), which defines the standard TIPS procedure. The investigators hypothesize that, in patients undergoing TIPS for the prevention of variceal rebleeding, stent underdilation using a 6-mm balloon (underdilated TIPS) will not increase the risk of rebleeding but may reduce the incidence of overt HE and attenuate liver injury. To test this hypothesis, the investigators have designed a prospective, multicenter, randomized controlled trial.

DETAILED DESCRIPTION:
Transjugular intrahepatic portosystemic shunt (TIPS) is a pivotal intervention for managing complications of portal hypertension. However, its clinical utility is limited by the risk of post-procedural hepatic encephalopathy (HE).

The pathogenesis of post-TIPS HE involves two principal mechanisms: the diversion of portal venous blood flow away from the liver and a concurrent reduction in hepatic metabolic capacity. Following TIPS placement, portal venous blood is shunted directly into the systemic circulation, resulting in decreased functional hepatic perfusion. This hemodynamic alteration not only increases the risk of HE but may also exacerbate pre-existing hepatic dysfunction. Evidence suggests that stent diameter plays a critical role in determining shunt patency, efficacy of portal pressure reduction, and the incidence of HE. A stent that is too narrow may inadequately lower portal pressure, leading to suboptimal therapeutic outcomes and an increased risk of shunt stenosis. Conversely, an excessively large stent can substantially increase the risk of HE and further impair liver function. Therefore, identifying an optimal stent diameter that effectively reduces portal pressure while minimizing complications-particularly shunt-induced HE-remains a central focus in TIPS research, aiming to balance procedural efficacy with safety to improve patient outcomes.

Early studies demonstrated that the use of stents with larger diameters than conventional calibers for the portal and hepatic veins was associated with a disproportionately increased risk of hepatic encephalopathy (HE) without substantial additional benefit in portal pressure reduction. Consequently, a stent diameter of 10 mm became the standard during the era of bare metal stents. However, the introduction of polytetrafluoroethylene (PTFE)-covered stents has significantly reduced the incidence of shunt dysfunction and improved the durability of portal pressure reduction following transjugular intrahepatic portosystemic shunt (TIPS) placement. Clinical evidence indicates that 8 mm PTFE-covered stents can maintain long-term patency and achieve adequate portal decompression while substantially lowering the risk of HE. Despite these advancements, the overall incidence of post-TIPS HE remains high, approximately 30%. To further optimize clinical outcomes, recent studies have explored a "stent underdilation" strategy, involving dilation of an 8 mm PTFE-covered stent using a 6 mm balloon. Preliminary data suggest that this approach may further reduce the incidence of HE without significantly increasing the risk of recurrent portal hypertensive events. Nevertheless, there is currently a lack of prospective, head-to-head randomized controlled trials comparing the efficacy and safety of underdilated TIPS versus standard-diameter TIPS in the management of complications related to portal hypertension.

In the context of managing gastroesophageal variceal bleeding, the established therapeutic goal of TIPS is to reduce the portosystemic pressure gradient (PPG) to less than 12 mmHg (16 cmH₂O). Building upon this principle, the investigators propose the following hypothesis: in patients with esophagogastric variceal bleeding undergoing TIPS, underdilated TIPS will reduce the incidence of overt HE and attenuate liver function deterioration without increasing the risk of rebleeding. To evaluate this hypothesis, the investigators have designed the present prospective clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years;
2. Diagnosis of liver cirrhosis based on clinical and imaging findings according to the 2023 Consensus Opinion on the Clinical Diagnosis and Treatment of Liver Cirrhosis in China (Chinese Society of Gastroenterology); histological confirmation required if diagnosis is inconclusive;
3. High-risk acute variceal bleeding, defined as presence of any of the following: Child-Pugh class C; Child-Pugh class B with active endoscopic evidence of bleeding; early rebleeding within 5 days; or failure of pharmacologic and endoscopic therapy to control bleeding;
4. History of esophagogastric variceal bleeding with documented failure of standard first-line therapy (endoscopic intervention plus nonselective beta-blocker, NSBB);
5. Scheduled to undergo TIPS;
6. Hepatic and renal function meeting all of the following criteria: Child-Pugh score ≤13; AST and ALT <5× upper limit of normal (ULN); serum creatinine <1.5× ULN;
7. Ability and willingness to provide written informed consent.

Exclusion Criteria:

(1) Budd-Chiari syndrome or other causes of non-cirrhotic portal hypertension; (2) current or prior malignancy, including hepatocellular carcinoma or extrahepatic malignancies; (3) complete thrombosis of the main portal vein; (4) severe psychiatric or neurological disorders (e.g., uncontrolled epilepsy, dementia); (5) history of liver resection or liver transplantation; (6) prior TIPS or surgical portosystemic shunt; (7) pregnancy or lactation; (8) any contraindication to TIPS, including severe right or left ventricular dysfunction, moderate-to-severe pulmonary hypertension despite optimal medical therapy, untreated severe valvular heart disease, or uncontrolled systemic infection; (9) acute variceal hemorrhage with MELD score ≥30 and/or arterial lactate >12 mmol/L, or presentation with acute-on-chronic liver failure (ACLF); (10) severe or refractory overt hepatic encephalopathy in the absence of a correctable spontaneous portosystemic shunt; (11) systemic conditions requiring ongoing systemic treatment with glucocorticoids or nonsteroidal anti-inflammatory drugs (NSAIDs).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of gastroesophageal variceal rebleeding. | Throughout the entire follow-up period（up to 12 months）
  Clinically significant rebleeding is defined in accordance with the Baveno V consensus criteria and is identified by recurrence of melena or hematemesis accompanied by any of the following: a) requirement for hospitalization; b) need for blood transfusion; c) hemoglobin decrease of ≥3 g/dL; or d) death within 6 weeks.

SECONDARY OUTCOMES:
All-cause rebleeding | Throughout the entire follow-up period（up to 12 months）
Stent dysfunction | 12 months
  Diagnosis of TIPS stent dysfunction follows a stepwise approach utilizing Doppler ultrasound, angiography, and measurement of the portosystemic pressure gradient (PPG). Stent dysfunction is diagnosed if either of the following criteria is met: (1) shunt stenosis ≥50% or complete occlusion; (2) an increase in PPG ≥25% compared to the baseline value measured immediately after stent placement. Angiography is indicated under the following circumstances: (1) recurrence of portal hypertension-related complications-TIPS stent dysfunction should be suspected upon recurrence of symptoms such as rebleeding, new-onset ascites, or persistence of ascites beyond 4-8 weeks; (2) color Doppler ultrasound findings-when flow direction is hepatofugal and mean maximum portal vein flow velocity (mVPmax) < 28 cm/s; when flow direction is hepatopetal and mVPmax < 39 cm/s.
New or worsening ascites | 12 months
  Defined as an increase of at least one grade in ascites severity on ultrasound (grading criteria: Grade 0 = none, Grade 1 = mild, Grade 2 = moderate, Grade 3 = large), or persistent ascites requiring paracentesis.
Incidence of overt hepatic encephalopathy | 12 months
  Hepatic encephalopathy is classified according to the 2022 European Association for the Study of the Liver (EASL) Clinical Practice Guidelines using the West-Haven criteria. Overt hepatic encephalopathy is defined as grade II or higher.
Liver function | 12 months
  Liver function will be evaluated using the Child-Pugh score (based on bilirubin, albumin, INR, ascites, and hepatic encephalopathy) and the Model for End-Stage Liver Disease (MELD) score.
Liver transplantation-free survival | 12 months
  Defined as the time from the TIPS procedure to the end of follow-up, liver transplantation, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Tie, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes